CLINICAL TRIAL: NCT02021032
Title: Post-Marketing Study Using PROLIEVE® for the Treatment of Benign Prostatic Hyperplasia (BPH)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medifocus, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101-04-401-01; NCT00407953 (obsolete NCT alias)
Record Dates: First submitted 2013-12-16; First posted 2013-12-27 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Benign Prostate Hyperplasia
Keywords: BPH
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prolieve (Experimental): Prolieve® is a transurethral microwave therapy device equipped with automated controls designed to deliver microwave energy to the prostate and balloon-administered compression for the treatment of symptomatic BPH. This device utilizes a transurethral catheter with microwave antenna to heat the prostate, with simultaneous 46 Fr. prostatic urethral catheter balloon-administered compression.
  Interventions: Device: Prolieve

INTERVENTIONS:
Device: Prolieve — Prolieve® is a transurethral microwave therapy device equipped with automated controls designed to deliver microwave energy to the prostate and balloon-administered compression for the treatment of symptomatic BPH. This device utilizes a transurethral catheter with microwave antenna to heat the prostate, with simultaneous 46 Fr. prostatic urethral catheter balloon-administered compression.

SUMMARY:
The primary objective of the post-marketing study is to collect safety and effectiveness data for 5 years on subjects treated with Prolieve®. The collection of 5-year safety information will be used to evaluate the occurrence of any long-term side effects from the treatment. The collection of long-term effectiveness data on subjects treated with Prolieve® will provide information on the long-term effects of treatment and time to re- treatment (any treatment initiated for BPH since Prolieve'" treatment, including a second treatment with Prolieve").

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with symptomatic BPH.
* Peak Urine flow rate <12 ml/sec on voided volume of >125mL.
* AUA symptom score value ≥9(9).
* Signed informed consent.

Exclusion Criteria:

* Subjects whose pain response has been significantly decreased by any means (because the subject's ability to detect pain is a treatment safety mechanism).
* Subject with a history of any illness or surgery that might confound the results of the study " or impede the successful completion of trial"
* Subject with a history of any illness for which the Prolieve® treatment may pose additional risk to the subject.
* Subject with the confirmed or suspected malignancy of the prostate
* Subject with the confirmed or suspected bladder cancer
* PSA >10 ng/mL
* Subject with previous treatment to the prostate (e.g., surgery, balloon dilation, stents, laser, TUNA, or Indigo prostatectomy) and/or non-metallic urogenital implants (e.g., penile prostheses, artificial urinary sphincters)
* Subject with prostate weighing <20 or >80g.
* Subject with previous pelvic irradiation or radial pelvic surgery
* Subject having large, obstructive middle lobe
* Previous rectal surgery (other than hemorrhoidectomy) or history of rectal disease.
* Subject with urethral stricture and/or bladder stones
* Active urinary tract infection.
* Subject with neurogenic bladder and/or sphincter abnormalities due to Parkinson's, multiple sclerosis, cerebrovascular accident (CVA), diabetes, or other disease process.
* Residual bladder volume >250 mL measured by ultrasound.
* Compromised renal function (i.e., serum creatinine levels above 1.8 mg/dL).
* Cardiac pacemaker or metallic implants or staples, etc. in the pelvic or femoral area.
* Concomitant medicating of the following:

  1. Bladder antispasmodics (Ditropan or Detrol) within one week of treatment, unless there is documented evidence that the subject has been on the same drug dose for at least three months with a stable voiding pattern. The drug dose will not be altered or discontinued for the entrance into or throughout the study.
  2. 5-alpha reductase inhibitors and gonadotropin releasing hormonal analog.
  3. Alpha blockers, antidepressants, androgens, within one week of treatment.
* Subject interested in future fertility/fathering children.
* Subject with full urinary retention.
* Subject with bleeding disorder or liver dysfunction associated with a bleeding disorder.
* Subject with prostatic urethra length of <1.2 cm or >5.5 cm.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2006-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Time to Re-Treatment | 5 years
  Time to re-treatment will be estimated using Kaplan Meier estimation techniques. The re-treatment rate at years 1 through 5 will be estimated and 95% confidence intervals obtained, and the median time to re-treatment will be estimated. Subjects who receive re-treatment will be classed as treatment failures. Subjects who are lost to follow-up will be considered as re-treated at their last known study visit. In addition, a missing at random (MAR) analysis will be performed.

SECONDARY OUTCOMES:
Change from Baseline in American Urological Association (AUA) Total Score at 5 years | 5 years
  Measured based on the number of subjects who worsened, had no change (1-29%), had a 30% or greater improvement or who are missing, based on the change in AUA total score compared to individual baseline for each follow-up evaluation. A responder analysis will also be done on peak flow rate (PFR) with the following categories: the number of subjects who worsened, had no change (1-19%), had a 20% or greater improvement or who are missing, based on the change in PFR compared to individual baseline for each follow-up evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Perry Weiner, MD, Study Director — Jefferson Urology
Locations (7):
- United States (7):
  - Winter Park Urology, Orlando, Florida
  - North Fulton Urology, Roswell, Georgia
  - Regional Urology, Shreveport, Louisiana
  - Merrimack Urology Associates PC, Chelmsford, Massachusetts
  - Albany Medical College Division of Urology, Alabany, New York
  - Midtown Urologic Trials, PC, New York, New York
  - Mobley Research Center, Houston, Texas

REFERENCES:
- [Derived] Olweny EO, Jow SL, Jow WW. Prolieve Transurethral Thermodilatation for Treatment of Symptomatic Benign Prostatic Hyperplasia: 5-Year Results from a Prospective Multicenter Trial. J Endourol. 2022 Jan;36(1):117-123. doi: 10.1089/end.2021.0240. Epub 2021 Nov 1. PMID 34314241